CLINICAL TRIAL: NCT05389176
Title: Effects of Heart Control at Different Stages on Hemodynamics Parameters and Clinical Prognosis in Patients of Septic Shock With Tachycardia
Brief Title: Effects of Heart Control at Different Stages in Patients of Septic Shock With Tachycardia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-038-02
Record Dates: First submitted 2022-04-28; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-03

CONDITIONS: Septic Shock; Tachycardia
Keywords: Septic Shock; Tachycardia; β receptor blockers
MeSH Terms: conditions — Shock, Septic; Tachycardia | interventions — esmolol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Esmolol is used 6 to 24 hours after onset of septic shock in patients with fluid optimization to control heart beats between 70-100bpm.
  Interventions: Drug: Esmolol
- Group B (Experimental): Esmolol is used 24 hours after onset of septic shock in patients to control heart beats between 70-100bpm.
  Interventions: Drug: Esmolol
- Group C (No Intervention): patients received conventional therapy in accordance with septic shock guidelines 2021

INTERVENTIONS:
Drug: Esmolol — a continuous esmolol infusion titrated to maintain heart rate between 70/min and 100/min
  Other Names: β-receptor blockers
  Arms: Group A; Group B

SUMMARY:
A sigle-center, randomized controlled trial will be do to investigate the effects of esomol on heart rate, clinical parameters, mortality, and safety in septic shock patients with tachycardia at different stages, compared with patients who received conventional therapy.

DETAILED DESCRIPTION:
The incidence of septic shock complicated with tachycardia is high and the prognosis is poor. Enough attention should be paid to and appropriate treatment should be given. High heart rate and high cardiac output are beneficial compensatory reactions of sepsis and septic shock. However, excessive sympathetic activation and high heart rate also have adverse effects on the cardiovascular system. Sustained tachycardia is harmful to patients with sepsis and septic shock and needs to be controlled. At present, it is widely used in the treatment of cardiovascular diseases and β Receptor blockers have the functions of preventing and reversing sympathetic effects, anti arrhythmia, anti-inflammatory and balancing myocardial oxygen supply and demand. Therefore, they are recommended to control arrhythmias in patients with septic shock. The 2014 guidelines for sepsis / septic shock in China suggest that if cardiac output is not low and the heart rate is fast after adequate fluid resuscitation, short acting drugs（β Receptor blockers）can be considered. However, there are some differences in the current clinical research results, and it suggests that the timing of treatment may affect the hemodynamic results and clinical outcomes of patients.

Therefore, this study intends to intervene with esmolol in patients with septic shock and tachycardia at different stages, and compare the hemodynamic parameters, clinical outcome, prognosis and adverse reactions with the conventional treatment group, in order to explore the appropriate time of esmolol in the treatment of patients with septic shock and tachycardia.

ELIGIBILITY:
Inclusion Criteria:

" ≥ 18 years old; " New septic shock within 24 hours, meeting the diagnostic criteria in 2012; " Septic shock lasts for more than 6 hours, and after fluid optimization using dynamic parameters, vasoactive drugs are still needed to maintain blood pressure; " the heart rate is greater than 100 beats / min for ≥ 1 hour，not caused by agitation, fever, and other factors; " informed consents are signed.

Exclusion Criteria:

" Shock caused by sepsis; " Septic cardiomyopathy or decreased myocardial contractility, requiring the use of positive inotropic drugs or significant cardiac insufficiency, such as CI ≤ 2.2l/min m2, PAWP>18mmHg, EF<40%; " Severe bronchial asthma or COPD; " Pregnant or lactating women; " Sinus bradycardia, degree II and degree III heart block; " β-receptor blockers were used before enrollment or have the history of sinus tachycardia; " Severe valvular heart disease; " Allergic to esmolol; " Tachycardia due to elevated body temperature, agitation, insufficient capacity and other reasons; " Have participated in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with heart rate of 70-100 bpm | at 24-hour after randomization
  the proportion of patients with heart rate of 70-100 bpm
the proportion of patients with heart rate of 70-100 bpm | at 48-hour after randomization
  the proportion of patients with heart rate of 70-100 bpm
the proportion of patients with heart rate of 70-100 bpm | at 72-hour after randomization
  the proportion of patients with heart rate of 70-100 bpm
the proportion of patients with heart rate of 70-100 bpm | at 96-hour after randomization
  the proportion of patients with heart rate of 70-100 bpm

SECONDARY OUTCOMES:
cardiac index | at 24-hour after randomization
  PiCCO monitoring parameters
cardiac index | at 48-hour after randomization
  PiCCO monitoring parameters
cardiac index | at 72-hour after randomization
  PiCCO monitoring parameters
cardiac index | at 96-hour after randomization
  PiCCO monitoring parameters
ejection fraction | at 24-hour after randomization
  cardiac measurement by cardiac ultrasound
ejection fraction | at 48-hour after randomization
  cardiac measurement by cardiac ultrasound
ejection fraction | at 72-hour after randomization
  cardiac measurement by cardiac ultrasound
ejection fraction | at 96-hour after randomization
  cardiac measurement by cardiac ultrasound
Arterial blood PH value | at 24-hour after randomization
  Arterial blood PH value by arterial blood gas analysis
Arterial blood PH value | at 48-hour after randomization
  Arterial blood PH value by arterial blood gas analysis
Arterial blood PH value | at 72-hour after randomization
  Arterial blood PH value by arterial blood gas analysis
Arterial blood PH value | at 96-hour after randomization
  Arterial blood PH value by arterial blood gas analysis
Arterial blood lactate | at 24-hour after randomization
  Arterial blood lactate by arterial blood gas analysis
Arterial blood lactate | at 48-hour after randomization
  Arterial blood lactate by arterial blood gas analysis
Arterial blood lactate | at 72-hour after randomization
  Arterial blood lactate by arterial blood gas analysis
Arterial blood lactate | at 96-hour after randomization
  Arterial blood lactate by arterial blood gas analysis
APACHEII scores | at 24-hour after randomization
  the Acute Physiology and Chronic Health Evaluation II scores，value 0～60, the higher score means worse outcome.
APACHEII scores | at 48-hour after randomization
  the Acute Physiology and Chronic Health Evaluation II scores，value 0~60, the higher score means worse outcome.
APACHEII scores | at 72-hour after randomization
  the Acute Physiology and Chronic Health Evaluation II scores，value 0~60, the higher score means worse outcome.
APACHEII scores | at 96-hour after randomization
  the Acute Physiology and Chronic Health Evaluation II scores，value 0~60, the higher score means worse outcome.
SOFA scores | at 24-hour after randomization
  sepsis-related organ failure assessment score，value 4~24, the higher score means worse outcome.
SOFA scores | at 48-hour after randomization
  sepsis-related organ failure assessment score，value 4~24, the higher score means worse outcome.
SOFA scores | at 72-hour after randomization
  sepsis-related organ failure assessment score，value 4~24, the higher score means worse outcome.
SOFA scores | at 96-hour after randomization
  sepsis-related organ failure assessment score，value 4~24, the higher score means worse outcome.
norepinephrine dose | at 24-hour after randomization
  norepinephrine dose (ug/kg.min)
norepinephrine dose | at 48-hour after randomization
  norepinephrine dose (ug/kg.min)
norepinephrine dose | at 72-hour after randomization
  norepinephrine dose (ug/kg.min)
norepinephrine dose | at 96-hour after randomization
  norepinephrine dose (ug/kg.min)
ICU- free days (by 28 days) | from randomization until 28 days
  days free of ICU
28-day mortality | from randomization until 28 days
  28-day mortality
days of mechanical ventilation | from randomization until 28 days
  days of mechanical ventilation
the incidence of hypotension deteriorated | by 96-hour after randomization
  the incidence of hypotension deteriorated
the incidence of heart arrest | by 96-hour after randomization
  the incidence of heart arrest

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, MD, Study Chair — The Affliated Drum Tower Hospital, Medical School of Nanjing University